CLINICAL TRIAL: NCT05173818
Title: Effect of Hyperbaric Oxygen on Persistent Post-concussive Symptoms After Mild Traumatic Brain Injury
Brief Title: Hyperbaric Oxygen Effects on Persistent Post-concussive Symptoms
Acronym: HOINPCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Essentia Health (Other)
Collaborators: University of North Dakota (Other); Dakota Medical Foundation (Unknown); The Swanson Foundation (Unknown); State of North Dakota (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EH21714
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Persistent Post-concussive Syndrome; Concussion Post Syndrome
Keywords: Hyperbaric oxygen treatment; Neurofilament light chain; RBANS
MeSH Terms: conditions — Post-Concussion Syndrome; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HBO at 1.5 Atmosphere absolute (Experimental): Participants in this group will be exposed to hyperbaric oxygen at 1.5 atmosphere absolute (ATA) for 60 minutes per session. Each participant will complete 40 sessions, five sessions per week within 3 months from randomization
  Interventions: Drug: Hyperbaric oxygen at 1.5 ATA
- Sham control initially at 1.2 then changed to 1.0 ATA (Sham Comparator): Participants in this group will be exposed to hyperbaric oxygen at 1.2 atmosphere absolute (ATA) during the first 5 to 7 minutes and the chamber pressure will be reduced to 1.0 ATA for the remaining 53 - 57 minutes for a total of 60 minutes per session. Each participant will complete 40 sessions, five sessions per week within 3 months from randomization
  Interventions: Drug: Sham treatment

INTERVENTIONS:
Drug: Hyperbaric oxygen at 1.5 ATA — Hyperbaric oxygen (HBO2) at 1.5 ATA (active) group (hyperbaric oxygen-chamber compressed to 1.5 atmosphere absolute and breathing >99.9% oxygen). Each participant should complete 40 sessions, one session per day, five per week over the course of 3 months.
  Other Names: 1.5 ATA
  Arms: HBO at 1.5 Atmosphere absolute
Drug: Sham treatment — Sham treatment includes pressurizing the chamber to 1.2 ATA with air for 5 minutes with noise of circulating air, return the chamber to 1.0 ATA after 5-7 minutes and maintain it at that pressure for until the end of the treatment, with noise of circulating air. Internal control knobs will be concealed. Participants will be instructed to undergo intermittent ear clearing technique during the initial 5 minutes of "descent"
  Other Names: 1.2 ATA then changed to 1.0 ATA
  Arms: Sham control initially at 1.2 then changed to 1.0 ATA

SUMMARY:
Persistent post-concussive symptoms (PPCS) are a source of significant burden among a subset of patients with concussion with prevalence rates previously reported between 11 - 82% based on timing of assessment, diagnostic criteria, or population under study.

Examples of persistent post-concussion symptoms include balance problems, headaches, fatigue, poor concentration, forgetfulness, anxiety, irritability, and sleep disturbance. Few proposed therapies have proved successful in the management of persistent post-concussion symptoms following mild traumatic brain injury.

The investigators will explore hyperbaric oxygen administered in a randomized sham-controlled clinical trial as an effective and tolerable treatment in improving neuropsychological status among adult patients with persistent post-concussive symptoms.

The overall hypothesis to be evaluated is that hyperbaric oxygen improves neuropsychological status and a serum concussion biomarker associated with PPCS.

DETAILED DESCRIPTION:
This is a parallel, randomized, double-blinded and sham-controlled study. A total of 100 subjects will be randomly assigned to either an intervention arm: 50 participants exposed to > 99.9% oxygen at 1.5 atmosphere absolute for 60 minutes over 40 treatments or sham-treatment arm: 50 participants exposed to oxygen and pressure composition equivalent to breathing atmospheric air for 60 minutes over 40 treatments.

This study is designed to determine whether hyperbaric oxygen improves neuropsychological status and ameliorates symptoms in adults with persistent post-concussive symptoms (PPCS) following mild traumatic brain injury. It recruits from either military or civilian population; uses a validated screening tool - Repeatable battery for the assessment of neuropsychological status (RBANS)- used in dementia and other forms of brain injury not used hitherto, in previous randomized control trial that investigated the effectiveness of hyperbaric oxygen in the management of PPCS. It also includes a concssuon biomarker, as an objective secondary endpoint.

The study is based on repeated measure design. The study will describe and track changes in the outcomes of interest over time, and examine associations between measures within each participant and across certain participant characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a history of mild traumatic brain injury, specifically, persistent post-concussive symptoms after examination by a neuropsychologist or neurologist.
* Volunteers time from concussive incident (Mild traumatic brain injury) must be between 3 months - 5 years following head trauma incident
* TBI was caused by non-penetrating trauma
* Volunteers must have current complaints of TBI symptoms such as headache, dizziness, or cognitive or affective problems
* Volunteers must be 18-year-old or more
* Willing and able to provide informed consent
* Able to speak and read English, as primary language
* Agrees to provide blood samples for clinical lab tests
* Willing and committed to comply with research protocol and complete all outcome measures
* Able to equalize middle ear pressures or willing to undergo needle myringotomies if needed
* Willingness and committed to comply with study protocol outlined reproductive plan based on baseline reproductive status

Exclusion Criteria:

* Prior treatment with hyperbaric oxygen treatment
* Hyperbaric chamber inside attendant, professional, SCUBA diver (technical, commercial, operational/military or recreational)
* The investigators will exclude pregnant women from this study because potential fetal adverse reactions triggered by high oxygen partial pressures such as retrolenticular fibroplasia though careful review of human data are generally reassuring such as the use of hyperbaric oxygen to treat acute carbon monoxide poison in the pregnant patient.13
* Prisoners
* Minors
* Unable to protect airway or requires frequent suctioning
* Known or suspected peri-lymphatic fistula
* Presence of tracheostomy (due to limitations in auto-inflating the middle ear)
* Unable to participate fully in outcome assessments
* Unable to cooperate with hyperbaric oxygen treatments
* Unable to speak and read English, as primary language
* Not cooperating with instructions during hyperbaric oxygen treatments such as bringing contraband items into the chamber (such as fire lighter)
* Not competent to sign their own consent. Such potential participants will not have the capacity to participate in a full range of neurocognitive testing
* Pre-existing diagnosis of a psychotic disorder(s): schizophrenia, bipolar, dissociative disorder
* History of moderate or severe traumatic brain injury
* History of brain injury not of traumatic etiology such as stroke or drug-induced coma
* Verifiable diagnosis of learning disability. Other pre-existing cognitive issues may make it difficult for potential participants to fill out certain outcome assessments such as neurobehavioral symptomatic inventory. This could lead to measurement bias or confound the result.
* Claustrophobia and unwilling to enter hyperbaric chamber
* Untreated pneumothorax
* Presence of implanted device with un-verifiable test to pressure by manufacturer
* Concurrent enrollment in an alternate interventional trial for post concussive symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in Repeatable battery for the assessment of neuropsychological status (RBANS) | Baseline, 1-week, 13-week, 18-month
  This is a validated screening tool initially used to assess dementia but has been extended to other neuropsychological conditions, including mild traumatic brain injury. RBANS can assess a broad range of independent neuropsychological domains, a characteristic of mild traumatic brain injury (affects different domains such as sleep, cognition). Alternate forms of RBANS allow for repeated evaluation and sensitivity to milder brain impairment.

SECONDARY OUTCOMES:
Changes in serum Neurofilament Light chain (NfL) level | Baseline, 1-week, 13-week, 18-month
  This is a protein marker of neuro-axonal damage that can be measured in serum and CSF. serum NfL has better diagnostic and prognostic utility than other neuro-axonal damage biomarkers such as GFAP, tau, UCH-LI in patients with TBI. There is Class III evidence that it distinguishes patients with mild TBI from healthy controls.
Changes in Pittsburg Sleep Quality Index (PSQI) score | Baseline, 1-week, 13-week, 18-month
  A validated self-rated subjective questionnaire comprising 19 individual questions that generate seven "component" scores {sleep quality, latency, duration, efficiency, disturbances, use of sleep medication and daytime dysfunction}. Persistent post-concussive symptoms following mild TBI usually affects several domains and patients could present with sleep disturbances, cognitive deficits, headache, dizziness, and behavioral changes.
  The 19 self-rated items are combined to form seven component scores; each of which has a range of 0-3 points. (0 = no difficulty, 3 = severe difficulty) and total score ranging from 0 - 21 points. "0" indicating no difficulty and "21" indicating severe difficulty in all areas. Higher scores indicate worse sleep quality
Changes in Neurobehavioral Symptom Inventory (NSI) scores | Baseline, 1-week, 13-week, 18-month
  This is a validated self-report measure of post-concussion symptoms, grouped into 4 cluster (somatosensory, cognitive, affective and vestibular).
  Neurobehavioral Symptom Inventor (NSI) is a 22 item symptoms scale, participants will rate the severity of their symptoms in the last 2 weeks on a 5 point likert scale (0=none, 1= mild, 2=moderate, 3=severe, 4=very severe) The NSI total score is a sum of the 22 items (range 0-88). Higher scores indicate more severe symptoms.
Changes in reported PTSD-Civilian version (PCL-C) measures | Baseline, 1-week, 13-week, 18-month
  This is a 17-item validated self-report measure that assesses PTSD symptoms. It is further subcategorized into three clusters (reexperiencing, avoidance, hyperarousal). A total score and cluster scores can be obtained based on DSM-IV-TR criteria.
  Participants rate how much they were "bothered by that problem in the past month". Items are rated on a 5-point scale ranging from 1 ("not at all") to 5 ("extremely"). A total score for the PTSD CheckList - Civilian Version (PCL-C) ranges from 17 - 85, and can be obtained by summing the scores from each of the 17 items. Higher scores indicate severe PTSD symptomatology.
Changes in World Health Organization Quality of Life -BREF (WHOQOL-BREF) domain scores | Baseline, 1-week, 13-week, 18-month
  World Health Organization Quality of Life - BREF is a practical abridged version of WHOQOL-100 that includes 26-item grouped into four domains (physical health, psychological, social relationships, environment). WHOQOL-100 has been shown to have good psychometric properties.
  WHOQOL-BREF creates a quality of life profile. Two items are examined separately. The other questions are grouped into four domains, and each domain score denote the participant's perception of quality of life in the index domain. The mean score of items within each domain is used to calculate the domain score. Mean scores are then multiplied by 4 in order to make domain scores comparable with the scores used in the WHOQOL-100. Higher domain scores denote higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Olayinka D Ajayi, MD, MPH, Principal Investigator — Essentia Health; Marc Basson, MD, PhD, Principal Investigator — University of North Dakota; Marilyn Klug, PhD, Study Chair — University of North Dakota; Paulina Kunecka, MD, Study Chair — Essentia Health; Richard Ferraro, PhD, Study Chair — University of North Dakota; Rebecca Quinn, MSW, LMSW, Study Chair — Center for Rural Health, University of North Dakota; Sharon Hanson, RN, Study Director — Essentia Health
Locations (1):
- Essentia Health, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical plan and consent form will be available on request. Data will be available on aggregate level; data will be deidentified, the full dataset and statistical code will be available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after study completion and for 36 months
Access Criteria: A full description of the intended use of the data must be sent to the corresponding author for review and approval. Participant consent for data sharing is conditioned and new ethics approval may be required.

REFERENCES:
- [Background] Moser RS, Schatz P. Enduring effects of concussion in youth athletes. Arch Clin Neuropsychol. 2002 Jan;17(1):91-100. PMID 14589756
- [Background] Shahim P, Politis A, van der Merwe A, Moore B, Chou YY, Pham DL, Butman JA, Diaz-Arrastia R, Gill JM, Brody DL, Zetterberg H, Blennow K, Chan L. Neurofilament light as a biomarker in traumatic brain injury. Neurology. 2020 Aug 11;95(6):e610-e622. doi: 10.1212/WNL.0000000000009983. Epub 2020 Jul 8. PMID 32641538
- [Background] Cook PA, Johnson TM, Martin SG, Gehrman PR, Bhatnagar S, Gee JC. A Retrospective Study of Predictors of Return to Duty versus Medical Retirement in an Active Duty Military Population with Blast-Related Mild Traumatic Brain Injury. J Neurotrauma. 2018 Apr 15;35(8):991-1002. doi: 10.1089/neu.2017.5141. Epub 2018 Mar 1. PMID 29239267
- [Result] Weaver LK, Wilson SH, Lindblad AS, Churchill S, Deru K, Price RC, Williams CS, Orrison WW, Walker JM, Meehan A, Mirow S. Hyperbaric oxygen for post-concussive symptoms in United States military service members: a randomized clinical trial. Undersea Hyperb Med. 2018 Mar-Apr;45(2):129-156. PMID 29734566